CLINICAL TRIAL: NCT02742220
Title: Effects of Isometric Handgrip Training on Blood Pressure Reduction in Patients With Peripheral Artery Disease: A Randomized Clinical Trial
Brief Title: Isometric Handgrip Training on Blood Pressure of Peripheral Artery Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Raphael M. Ritti Dias, PhD, University of Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IHT PAD
Record Dates: First submitted 2016-04-04; First posted 2016-04-18 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Peripheral Artery Disease
Keywords: intermittent claudication; exercise; blood pressure; cardiovascular system
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isometric Handgrip Training Group (Experimental): Experimental group will perform home-based unilateral handgrip exercise and will be recommended to increase daily physical activity levels.
  Interventions: Other: Isometric Handgrip Training Group
- Control Group (Sham Comparator): Control group will be recommended to increase daily physical activity levels.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Isometric Handgrip Training Group — Intervention period will last eight weeks. Experimental group will perform three sessions per week of home-based handgrip exercise. The exercise protocol will consist of four unilateral sets (dominant arm) with two minutes of isometric contraction, with 30% of maximum voluntary contraction, and four minutes of interval between sets. Patients will receive a diary to record the sessions and report difficulties during the training. Visits will be scheduled at weeks 1 and 5 to provide feedback to individuals, discuss possible problems during the training and adjust the intensity of the exercise. In addition the patients be recommended to increase daily physical activity levels, and weekly, there will be phone contacts with the patients to reinforce the exercise recommendations.
  Other Names: Isometric resistance exercise
  Arms: Isometric Handgrip Training Group
Other: Control Group — Intervention period will last eight weeks. Patients will be recommended to increase daily physical activity levels, and weekly, there will be phone contacts to reinforce the recommendations.
  Arms: Control Group

SUMMARY:
The aim of this study is to analyze the effects of isometric handgrip training (IHT) on blood pressure of hypertensive patients with peripheral arterial disease. Will be recruited 60 patients which will be randomized into 2 groups (30 per group), IHT and control group (CG). IHT group will training isometric contraction for 8 weeks. The GC patients will be encouraged to increase the level of physical activity. In the pre and post-intervention, brachial and central blood pressure will be measured.

DETAILED DESCRIPTION:
Meta-analyze studies have shown that IHT promotes reductions in blood pressure (BP), reaching 10 mmHg for systolic and diastolic 7 mmHg. However, remain uncertain the effects of this type of training on BP in patients with more severe cardiovascular diseases such as peripheral artery disease. Because this type of training which requires approximately 20 minutes per session and does not require supervision, it is possible that this intervention is interesting to reduce BP of these patients. The aim of this study is to analyze the effects of IHT on blood pressure of hypertensive patients with peripheral arterial disease. Will be recruited 60 patients, which will be randomized into 2 groups (30 per group), IHT and control group (CG). IHT group will hold three sessions per week with four unilateral sets with two minutes of isometric contraction at 30% of maximal voluntary contraction and interval of four minutes between them, for 8 weeks. The GC patients will be encouraged to increase the level of physical activity. In the pre and post-intervention, is going to be evaluated functional capacity, brachial and central BP, arterial stiffness, cardiovascular autonomic modulation and muscle vasodilation. Will be used to analyze two-factor variance for repeated measures, with group (IHT and GC) and the time (before and after 8 weeks) as factors and the post-hoc test of Newman-Keuls.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal without hormone therapy replacement, if woman;
* present peripheral artery disease (ankle brachial index < 0.90) in one or both lower limbs;
* do not present neurological / cognitive diseases;
* is able to practice home-based exercise;

Exclusion Criteria:

* patients will only be excluded if they make any medication changes before completing the intervention period or present any health problems that prevent physical activity.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood pressure at eight weeks | Baseline and eight weeks
  Blood pressure will be measured before and after eight weeks of intervention period on intervention and control group by an automatic blood pressure monitor (HEM-742, Omron Healthcare, Japan).

SECONDARY OUTCOMES:
Change from baseline in autonomic cardiac modulation at eight weeks | Baseline and eight weeks
  Cardiac autonomic modulation will be measured before and after eight weeks of intervention period on intervention and control group by heart rate monitor (Polar, RS 800, USA).
Change from baseline in vasodilatory capacity at eight weeks | Baseline and eight weeks
  Vasodilatory capacity will be measured before and after eight weeks of intervention period on intervention and control group by a flow mediated dilation measurement with an ultrasound image (HDI 5000 Sono CT, Philips, The Netherlands).
Change from baseline in arterial stiffness at eight weeks | Baseline and eight weeks
  Arterial stiffness will be measured before and after eight weeks of intervention period on intervention and control group by pulse wave velocity measurement with applanation tonometry (SphygmoCor, AtCor Medical, Australia).

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Ritti-Dias, PhD, Principal Investigator — Israel Institute of Education and Research Albert Einstein; Gabriel Cucato, PhD, Study Director — Israel Institute of Education and Research Albert Einstein
Locations (1):
- Israel Institute of Education and Research Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The IPD data to be shared are the indivividual and mean data of blood pressure responses to eight weeks of isometric handgrip training.

REFERENCES:
- [Derived] A Correia M, Oliveira PL, Farah BQ, Vianna LC, Wolosker N, Puech-Leao P, Green DJ, Cucato GG, Ritti-Dias RM. Effects of Isometric Handgrip Training in Patients With Peripheral Artery Disease: A Randomized Controlled Trial. J Am Heart Assoc. 2020 Feb 18;9(4):e013596. doi: 10.1161/JAHA.119.013596. Epub 2020 Feb 6. PMID 32067595